CLINICAL TRIAL: NCT01291576
Title: Randomized Trial Comparing Digestive and Urinary Dysfunction Secondary to 2 Surgical Techniques Used in the Management of Deep Endometriosis Infiltrating the Rectum: Colorectal Resection and Rectal Nodules Excision (ENDORE)
Brief Title: Functional Outcomes of Surgical Management of Deep Endometriosis Infiltrating the Rectum
Acronym: ENDORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2009/069/HP
Record Dates: First submitted 2011-01-31; First posted 2011-02-08 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Endometriosis, Rectum
Keywords: Deep infiltrating endometriosis; Rectal endometriosis; Colorectal resection; Nodule excision; Rectal shaving; Functional outcomes; Constipation
MeSH Terms: conditions — Endometriosis; Constipation | interventions — Administration, Rectal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectal/colorectal segmental resection (Active Comparator)
  Interventions: Procedure: Rectal/colorectal segmental resection
- Rectal nodule excision (Active Comparator)
  Interventions: Procedure: Rectal nodule excision

INTERVENTIONS:
Procedure: Rectal/colorectal segmental resection — Resection of the rectum +/- sigmoid colon involved by the deep infiltrating endometriosis
  Other Names: Anterior rectal resection
  Arms: Rectal/colorectal segmental resection
Procedure: Rectal nodule excision — Either full thickness excision or rectal shaving
  Other Names: Conservative sergery of the rectum
  Arms: Rectal nodule excision

SUMMARY:
The purpose of this study is to determine whether performing colorectal resection in deep endometriosis infiltrating the rectum is responsible for a higher rate of postoperative digestive and urinary dysfunction when compared to rectal nodules excision (conservation of the rectum).

DETAILED DESCRIPTION:
The study compare digestive and urinary functional outcomes following surgical management of rectal endometriosis by either colorectal resection or conservative surgery (shaving or full thickness excision of rectal nodules).

Patients managed for rectal endometriosis are randomized in two arms, and followed up for 24 months. The assessment of digestive and urinary functions is performed at 6, 12, 18 and 24 months using standardized questionnaires. Postoperative complications and improvement of endometriosis related pain are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* female
* age >18 and <45
* at least one digestive symptom related to deep endometriosis (pain defecation, either cyclic diarrhea or cyclic constipation, cyclic rectorrhagia)
* preoperative work up revealing a deep endometriosis nodule infiltrating the rectum (either muscular or submucosal layer, on less than 50% of rectal circumference) and measuring at least 20 mm
* affiliation to the National Social Security System

Exclusion Criteria:

* pregnant women or likely to be at the moment of the surgery
* no preoperative hypothesis of rectal involvement
* no intraoperative confirmation of the rectal involvement
* advanced rectal endometriosis involving rectal mucosa or more than 50% of the rectal circumference (preoperative assessment using rectal endoscopy or ultrasonography)
* women unable to give an informed consent (guardianship or trusteeship)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
Percentage of women experiencing a postoperative digestive or urinary dysfunction | 24 months
  At least one of following symptoms:
  * major constipation (< 1 stool/5 days) associated with defecation pain;
  * increase of the stool frequency ( >=3 stools/day);
  * anal incontinence;
  * de novo postoperative dysuria confirmed by urodynamic work up;
  * bladder atony requiring daily catheterization.

SECONDARY OUTCOMES:
Percentage of women experiencing postoperative pain related to endometriosis | 24 months
  Percentage of women presenting with dysmenorrhea, dyspareunia, chronic pelvic pain
Percentage of women experiencing a postoperative digestive or urinary dysfunction | 12 months
  At least one of following symptoms:
  * major constipation (< 1 stool/5 days) associated with defecation pain;
  * increase of the stool frequency ( >=3 stools/day);
  * anal incontinence;
  * de novo postoperative dysuria confirmed by urodynamic work up;
  * bladder atony requiring daily catheterization.
Biberoglu & Behrman score | 24 months
  Evaluation of endometriosis related pain using the above mentioned scale
SF-36 quality of life scale | 24 months
The Gastrointestinal Quality of Life Index (GIQLI) | 24 months
The Knowles-Eccersley-Scott-Symptom Questionnaire (KESS) | 24 months
Wexner questionnaire related to anal incontinence | 24 months
percentage of women requiring endoscopic dilatation due to the stenosis of the colorectal anastomosis | 24 months
Percentage of women presenting postoperative rectal fistulae or leakage of rectal suture or colorectal anastomosis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Horace Roman, MD PhD, Principal Investigator — Rouen University Hospital, France
Locations (3):
- France (3):
  - Service de Gynécologie et Obstétrique, CHU Jean de Flandre, Lille
  - Service de Gynécologique-Obstétricale et Reproduction Humaine, Hôpital Tenon, Université Pierre et Marie Curie Paris 6, Paris
  - Rouen University Hospital, Rouen

REFERENCES:
- [Derived] Roman H, Tuech JJ, Huet E, Bridoux V, Khalil H, Hennetier C, Bubenheim M, Branduse LA. Excision versus colorectal resection in deep endometriosis infiltrating the rectum: 5-year follow-up of patients enrolled in a randomized controlled trial. Hum Reprod. 2019 Dec 1;34(12):2362-2371. doi: 10.1093/humrep/dez217. PMID 31820806
- [Derived] Roman H, Chanavaz-Lacheray I, Ballester M, Bendifallah S, Touleimat S, Tuech JJ, Farella M, Merlot B. High postoperative fertility rate following surgical management of colorectal endometriosis. Hum Reprod. 2018 Sep 1;33(9):1669-1676. doi: 10.1093/humrep/dey146. PMID 30052994